CLINICAL TRIAL: NCT05307952
Title: Auditory Diagnostics and Error-based Treatment
Acronym: AuDiET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-13495
Record Dates: First submitted 2022-03-10; First posted 2022-04-01 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Deafness, Bilateral; Deafness Neurosensory; Deafness Permanent
Keywords: Cochlear Implant; Speech Perception; Hearing; Speech; Prosthesis Fitting; Rehabilitation
MeSH Terms: conditions — Hearing Loss, Bilateral; Hearing Loss, Sensorineural; Deafness; Speech | interventions — Audiometry, Pure-Tone; Speech Perception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fitting and Training Intervention (Experimental): All participants will undergo the full set of diagnostic visits and both Fitting and Training interventions.
  The Fitting Intervention is an adjustment of their processors' MAPs based on their error pattern.
  The Training Intervention is a personalized training via an app focusing on their most frequent errors.
  Interventions: Diagnostic Test: Tone Audiometry; Diagnostic Test: Spectrotemporal Assessment; Diagnostic Test: Phoneme and Speech Perception; Diagnostic Test: Digit Triplet Test; Other: Personalized fitting; Behavioral: Personalized training

INTERVENTIONS:
Diagnostic Test: Tone Audiometry — Evaluation of the participants' audiometrical thresholds
Diagnostic Test: Spectrotemporal Assessment — Evaluation of the participants' promptness in detecting a modulation of a harmonic complex
Diagnostic Test: Phoneme and Speech Perception — Evaluation of the participants' understanding of phonemes and short words, both in quiet and in noise
Diagnostic Test: Digit Triplet Test — Evaluation of the participants' ability to discern speech in noise
Other: Personalized fitting — Adjustment of the parameters of the participants' cochlear implants aimed at improving their speech perception
Behavioral: Personalized training — Self-administered training exercises focused on the speech components the participants are experiencing difficulties into

SUMMARY:
The main objective of this study is to assess the effectiveness of an integrated program of fitting and training interventions aimed at reducing unexpected variability and addressing the specific error patterns of each recipient.

The participants will undergo 1 visit lasting approximately 2 hours at the Radboud university medical center's ENT department, where they will undergo a series of diagnostic tests. Some of the participants will also be asked to self-administer additional tests using a Windows tablet.

Based on the outcomes of speech recognition tests in quiet at the first visit, the participants will be called for follow-up interventions concerning both the fitting of their CI and personalized auditory training based on their personal error patterns. These interventions will take place over the course of approximately 5 months and will be made up of three follow-up visits and a period of self-administered training through a mobile application on a tablet.

One final follow-up visit will check whether any changes from the interventions are retained after four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult (over 18 years old at the time of inclusion )
* Post-lingually deafened (the subject had a good mastery of spoken language before onset of deafness)
* Native Dutch speaker
* Implanted, either unilaterally or bilaterally, with a Cochlear Implant manufactured by Cochlear Ltd (i.e., a Nucleus ® implant).
* Implanted with one of the following implants: CI422, CI512, CI522, CI532, CI24M, CI24R, CI24RE.
* Implanted for at least 12 months.

Exclusion Criteria:

* Known abnormally formed cochlea
* Known pre-implantation ossification of the cochlea
* Severe cognitive disorders affecting their ability to understand spoken language
* Intense facial nerve stimulation
* Unaddressed electrode tip foldover
* More than 4 electrodes deactivated because of malfunction (open/short circuit) or lack of response
* Additional illnesses or handicaps that could impact ability to participate in study, at the clinician's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in Percent Speech Recognition | Weeks 1, 10, 14, 18
  Given a list of CNC words, this score measures the percentage of correctly identified words.

SECONDARY OUTCOMES:
Change in Distance-based Accuracy Score | Weeks 1, 10, 14, 18
  Speech Recognition accuracy score based on phoneme distance, such that mistaking a phoneme for a similar one such as mistaking /k/ for /g/ gives a lower penalty than mistaking a phoneme for a very different one.
Change in Error Dispersion | Weeks 1, 10, 14, 18
  Mathematical quantification of how much the errors made by the subjects are spread between stimuli and responses

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Huinck, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to any researchers not involved in the project

REFERENCES:
- [Derived] Philpott N, Philips B, Wasmann JW, Migliorini E, van Dijk B, Mylanus EAM, Huinck WJ. Individualized home-based phoneme training for adult cochlear implant users reduces phoneme confusion errors. Cochlear Implants Int. 2025 Sep;26(5):363-373. doi: 10.1080/14670100.2025.2583654. Epub 2025 Nov 11. PMID 41219176